CLINICAL TRIAL: NCT04698226
Title: Internal Limiting Membrane Peeling Versus Inverted Flap Technique for Treatment of Idiopathic Full-thickness Macular Hole: a Comparative Study of Near Visual Acuity Outcomes Using Salzburg Reading Desk.
Brief Title: ILM Peeling Versus Inverted Flap Technique for Treatment of Macular Hole: Near Visual Acuity Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Collaborators: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Martin Pencak, Principal Investigator, Faculty Hospital Kralovske Vinohrady
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH SRD V1.0
Record Dates: First submitted 2021-01-02; First posted 2021-01-06 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Macular Holes
Keywords: Idiopathic macular hole; Pars plana vitrectomy; Inverted flap; Internal limiting membrane peel; Salzburg reading desk; Microperimetry
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ILM peel (Active Comparator): Patients who will undergo 25-gauge pars plana vitrectomy with complete internal limiting membrane peeling and SF6 tamponade.
  Interventions: Procedure: 25-gauge pars plana vitrectomy with complete internal limiting membrane peeling and SF6 tamponade
- Inverted flap (Experimental): Patients who will undergo 25-gauge pars plana vitrectomy with inverted flap technique and SF6 tamponade.
  Interventions: Procedure: 25-gauge pars plana vitrectomy with inverted flap technique and SF6 tamponade

INTERVENTIONS:
Procedure: 25-gauge pars plana vitrectomy with complete internal limiting membrane peeling and SF6 tamponade — Standard 3 port 25-gauge pars plana vitrectomy with complete internal limiting membrane peeling around the macular hole after brilliant blue dye staining and sulfur hexafluoride (SF6) tamponade
  Arms: ILM peel
Procedure: 25-gauge pars plana vitrectomy with inverted flap technique and SF6 tamponade — Standard 3 port 25-gauge pars plana vitrectomy with inverted flap technique after brilliant blue dye staining and SF6 tamponade. "Flower petal" type of inverted flap will be performed - multiple small ILM flaps will be created around the macular hole and placed over the macular hole.
  Arms: Inverted flap

SUMMARY:
A prospective randomised study comparing the near visual acuity outcomes using Salzburg Reading Desk in pseudophakic patients with idiopathic full-thickness macular hole treated with pars plana vitrectomy with internal limiting membrane peeling versus inverted flap technique. The aim of the study is confirm or disprove the hypothesis, that the near visual acuity results of pars plana vitrectomy with inverted flap technique for idiopathic macular hole are not inferior to pars plana vitrectomy with complete internal limiting membrane peeling technique. Patients will be followed for 6 months after the operation and near best corrected visual acuity testing on Salzburg reading desk, distance best corrected visual acuity on ETDRS tables and microperimetry will be performed and compared between both groups. Also the macular hole closure rate and complication rate will be compared between both groups.

DETAILED DESCRIPTION:
Idiopathic full-thickness macular hole (MH) is an anatomic defect of the macula caused by the traction of the vitreous. Interruption of all neural retinal layers from the internal limiting membrane (ILM) to the retinal pigment epithelium (RPE) is present. Although other therapeutic approaches like pneumatic or enzymatic vitreolysis may lead to MH closure, pars plana vitrectomy (PPV) remains a gold standard for the treatment of full-thickness MH. Combination of PPV with full ILM peeling showed excellent results in small to medium MH, however the success rates dropped significantly with the increasing size of MH. PPV with inverted flap technique was introduced to address this issue and showed great results in MH of all diameters. In inverted flap technique, ILM is peeled around the MH and small piece of it is placed over the MH. It is speculated, that it serves as a scaffolding for gliosis allowing it to close large MHs. Besides gliosis, the ILM flap seals the MH by secluding communication between the vitreous and subretinal space, creating a closed compartment enabling the RPE to pump out fluid effectively. However, it is not known whether the ILM left in the macular hole might not hinder the healing process and full closure of macular hole. The aim of this study is to perform a detailed assessment of the state of the macula and near best corrected visual acuity and to compare the results of complete ILM peeling and ILM flap technique.

This is a prospective randomised study comparing the near visual acuity outcomes using Salzburg Reading Desk in pseudophakic patients with idiopathic full-thickness MH treated with PPV with ILM peeling versus inverted flap technique. Participants are randomized in a 1:1 ration to undergo 25-gauge PPV with complete ILM peeling or with circular inverted flap technique with sulphur hexafluoride as a tamponade and recommendation to maintain reading position for 3 days.

At baseline visit (D1) one day prior to the operation, patients undergo distance best corrected visual acuity (BCVA) exam using ETDRS charts, intraocular pressure (IOP) measuring using the non-contact tonometry, anterior segment slit-lamp examination, fundus biomicroscopy, microperimetry and optical coherence tomography (OCT).

At month 3 (M3) and month 6 (M6) visits, patients undergo distance BCVA exam using ETDRS charts, near BCVA exam using the Salzburg reading desk (SRD Vision, NY, USA), IOP measuring using the non-contact tonometry, anterior segment slit-lamp examination, fundus biomicroscopy, microperimetry, and OCT. The closure of macular hole and post-operational complications are assessed.

Distance BCVA is performed using ETDRS charts and recorded in logMAR.

Microperimetry is performed using the MAIA Confocal Microperimeter (CenterVue S.p.A, Padova, Italy). Expert exam 4-2 of the study eye is performed two times and the average of macular integrity score, average threshold score and fixation stability P1 and P2 are recorded.

OCT is performed using the Spectralis OCT (Heidelberg Engineering GmbH, Heidelberg, Germany). Macula of the study eye is scanned in 512 horizontal scans in the angle of 20x20 degrees with the spacing of 11 um in High Speed mode with noise reduction set to ART=5. The minimum and basal macular hole diameter is recorded, and the staging of the macular hole is performed using both the Gass and International Vitreomacular Traction Study Classification System. Presence or absence of epiretinal membrane is recorded.

Near BCVA is performed using the Salzburg reading desk. The best near correction is determined first using the Jaeger Reading Eye Charts. Examination on Salzburg reading desk is performed afterwards in Czech with the reading distance set to 40 cm with contrast and luminance set to 100%. Progressively smaller text is presented to the patient until his reading speed falls under 80 words per minute (wpm) or until his word miss rate is higher than 1. At this point, patient is presented with 5 different sentences with the same text size. Test is ended if the patient cannot exceed the reading speed of 80 wpm or if his word miss rate is higher than 1 3 or more times for the same text size. The smallest text size where reading speed is over 80 wpm or word miss rate is 1 or lower is recorded in logMAR as near BCVA.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age
* With idiopathic full thickness macular hole verified on OCT (Gass stage 2-4)
* Minimal macular hole size under 1000 um
* Pseudophakic

Exclusion Criteria:

* Presence of other ocular pathology influencing visual acuity (e.g. age-related macular degeneration, diabetic retinopathy etc.)
* Unwilling to sign the informed consent form
* Unable to come to the study visits
* Health status not allowing participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Near best corrected visual acuity on Salzburg reading desk | Month 6
  Near best corrected visual acuity defined as the smallest text size where reading speed is over 80 wpm or word miss rate is 1 or lower as per Salzburg reading desk exam.
Microperimetry - macular integrity | Baseline and month 6
  Change from baseline macular integrity score from MAIA Confocal Microperimeter Expert exam 4-2 of the study eye at month 6.
Microperimetry - avarage threshold | Baseline and month 6
  Change from baseline avarage threshold score from MAIA Confocal Microperimeter Expert exam 4-2 of the study eye.exam 4-2 of the study eye at month 6.
Microperimetry - fixation stability | Baseline and month 6
  Change from baseline fixation stability P1 and P2 from MAIA Confocal Microperimeter Expert exam 4-2 of the study eye at month 6.
Macular hole closure rate | Month 6
  Macular hole closure rate defined as a flattened and reattached hole rim along the whole circumference of macular hole on the OCT examination of the macular region of the study eye.

SECONDARY OUTCOMES:
Distance best corrected visual acuity | Baseline and month 6
  Change from baseline distance best corrected visual acuity examined on ETDRS tables and recorded in logMAR at month 6.
Occurrence of perioperative complications | Month 3
  Occurrence of perioperative complications such as retinal breaks, etc. will be recorded.
Occurrence of postoperative complications | Month 6
  Occurrence of postoperative complications such as intraocular haemorrhage, retinal detachment etc. will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Pencak, M.D., Principal Investigator — Faculty Hospital Kralovske Vinohrady
Locations (1):
- Department of Ophthalmology, Faculty hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No